CLINICAL TRIAL: NCT00583154
Title: A Pilot Efficacy Evaluation of BLI-801 as a Laxative in Constipated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Clinical Operations Manager, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLI-801-101
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Constipation
Keywords: constipation; laxative
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): BLI-801 Dose 1
  Interventions: Drug: BLI-801
- 2 (Experimental): BLI-801 Dose 2
  Interventions: Drug: BLI-801
- 3 (Experimental): BLI-801 Dose 3
  Interventions: Drug: BLI-801
- 4 (Experimental): BLI-801 Dose 4
  Interventions: Drug: BLI-801

INTERVENTIONS:
Drug: BLI-801 — Dose 1
  Arms: 1
Drug: BLI-801 — Dose 2
  Arms: 2
Drug: BLI-801 — Dose 3
  Arms: 3
Drug: BLI-801 — Dose 4
  Arms: 4

SUMMARY:
To compare the safety and efficacy of BLI-801 administered at 4 dose levels in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age
* Constipated according to ROME I criteria
* Otherwise in good health, as determined by physical exam and medical history
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse)
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
* Subjects taking laxatives or prokinetic agents that refuse to discontinue these treatments for the duration of the study
* Subjects who are pregnant or lactating, or intending to become pregnant during the study
* Subjects of childbearing potential who refuse a pregnancy test
* Subjects who are allergic to any BLI-801 component.
* Subjects who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Bowel Movement Count | 24 hours

SECONDARY OUTCOMES:
Adverse events | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (3):
- United States (3):
  - Anaheim, California
  - Cranston, Rhode Island
  - Cumberland, Rhode Island